CLINICAL TRIAL: NCT00817518
Title: An Open-label, Dose-escalation Study With Extension to Evaluate Safety, Pharmacokinetics and Anti-tumor Activity of RO4987655, a MEK Inhibitor, Administered Orally as Monotherapy in Patients With Advanced Tumors
Brief Title: A Dose-Escalating Study of RO4987655 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO21189; 2007-002021-77
Record Dates: First submitted 2008-12-16; First posted 2009-01-06 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-09

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — CH 4987655

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: RO4987655
- 2 (Experimental)
  Interventions: Drug: RO4987655

INTERVENTIONS:
Drug: RO4987655 — Administered po daily for 28 days, at escalating doses, with a starting dose of 1mg (Part 1) maximum tolerated dose administered po daily until disease progression(Part 2)
  Arms: 1
Drug: RO4987655 — Administered po daily for 28 days, at escalating doses , with a starting dose of 1mg (Part 1). Optimal biological dose administered po daily until disease progression (Part 2)
  Arms: 2

SUMMARY:
This study will determine the maximum tolerated dose and the dose-limiting toxicities of RO4987655 in patients with advanced and/or metastatic solid tumors. In the first part of the study, groups of patients will be sequentially enrolled to receive ascending oral doses of RO4987655 daily for 28 days. The starting dose of 1mg daily will be escalated in subsequent groups of patients after a successful assessment of the safety and tolerability of the previous dose. In Part 2 of the study, patients with metastatic or advanced malignant melanoma, or any other responsive tumor type, will be randomized to receive either the maximum tolerated dose or the optimal biological dose of RO4987655 daily. The anticipated time on study treatment is until disease progression, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* advanced and/or metastatic cancer not amenable to standard therapy;
* any solid tumor type (Part 1); malignant melanoma or other responsive tumor type (Part 2);
* measurable and/or evaluable disease (Part 1); >=1 measurable lesion (Part 2);
* ECOG performance status 0-2.

Exclusion Criteria:

* prior chemotherapy, radiotherapy or immunotherapy within 28 days of first receipt of study drug;
* prior corticosteroids as anti-cancer therapy within 14 days of first receipt of study drug;
* active CNS lesions;
* acute or chronic infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2009-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (Part 1) | Reviewed after each 4 week cycle
Tumor assessments (Part 2) | Every 8 weeks

SECONDARY OUTCOMES:
Adverse events, laboratory parameters, PD parameters, optimal biological dose (Parts 1 and 2) | Reviewed after each 4 week cycle

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (11):
- France (3):
  - Marseille
  - Paris
  - Villejuif
- Essen, Germany
- Amsterdam, Netherlands
- Spain (3):
  - Barcelona, Barcelona
  - Madrid, Madrid
  - Seville, Sevilla
- United Kingdom (3):
  - Cambridge
  - London
  - Oxford